CLINICAL TRIAL: NCT01530204
Title: RAPID: Reducing Pain; Preventing Depression
Acronym: RAPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jordan F. Karp, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MH090333 Sub-Project ID: 8317
Record Dates: First submitted 2012-02-01; First posted 2012-02-09 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee arthritis; knee osteoarthritis; knee pain; cognitive behavioral therapy; physical therapy; depression prevention
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Physical Therapy (Active Comparator): 8-12 sessions of knee-focused physical therapy and a home-based conditioning program.
  Interventions: Procedure: Physical Therapy for knee OA
- Cognitive Behavioral Therapy for Pain (Active Comparator): 8-12 session pain-focused Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy for Pain CBT-P
- Enhanced Treatment as Usual (Active Comparator): Information about state-of-the-art pharmacotherapy for osteoarthritis is communicated to the primary care physicians of participants.
  Interventions: Other: Enhanced Treatment as Usual

INTERVENTIONS:
Procedure: Physical Therapy for knee OA — 8-12 sessions of knee-focused physical therapy and a home-based conditioning program.
  Arms: Physical Therapy
Behavioral: Cognitive Behavioral Therapy for Pain CBT-P — 8-12 session pain-focused Cognitive Behavioral Therapy
  Arms: Cognitive Behavioral Therapy for Pain
Other: Enhanced Treatment as Usual — Information about state-of-the-art pharmacotherapy for osteoarthritis is communicated to the primary care physicians of participants.
  Arms: Enhanced Treatment as Usual

SUMMARY:
The primary question addressed by this prevention study is to explore if improving pain and disability reduces episodes of Major Depression among seniors with knee osteoarthritis (OA) and mild depressive symptoms.

DETAILED DESCRIPTION:
In this Sequential Multiple Assignment Randomized (SMART) Trial, the investigators care comparing Cognitive Behavioral Therapy for Pain (CBT-P) with EXERCISE (knee-specific Physical Therapy) delivered individually and sequentially. A subset of participants will receive enhanced care as usual in which their primary care physicians will receive information about pharmacological management of knee osteoarthritis. The active phase of the study may be up to 16 weeks, and the follow-up period lasts 12 months.

Stage 1, Specific Aim 1: To test if Cognitive Behavioral Therapy for Pain (CBT-P) results in more improvement in pain and disability than those receiving knee-specific Physical Therapy (EXERCISE).

Stage 1, Hypothesis 1: At week 8, subjects randomized to CBT-P will have more improvement in pain and disability than those randomized to EXERCISE.

Stage 2, Specific Aim 2: For non-responders to Stage 1, to explore which sequence of interventions leads to greater improvement in pain and disability.

Stage 2, Hypothesis 2: Compared to the other sequenced interventions (see Figure), subjects randomized to CBT-P and then EXERCISE will have the most improvement in pain and disability.

Follow-up, Specific Aim 3: To explore if improvement in pain and disability is associated with incident major depressive episode (MDE) over 12 months.

Follow-up, Hypothesis 3: More pain and disability improvement will be associated with lower rates of incident (MDE) over 12 months.

Exploratory AIM 1: To compare "legacy" assessments of functioning and psychological health with Computer Adaptive Testing (CAT) assessments of these domains for level of agreement.

Exploratory AIM 2: To assess candidate genetic polymorphisms, peripheral mRNA biosignatures, and candidate cytokine and growth factor levels using both multiplex assays and individual ELISAs. The investigators are exploring if these biomarkers are associated with pain improvement and risk for developing MDE.

ELIGIBILITY:
Inclusion Criteria:

1. >/= age 60
2. meets accepted clinical criteria for knee OA based on the American College of Rheumatology 1986 clinical criteria guidelines.
3. Western Ontario and McMaster University Arthritis Index (WOMAC) pain subscale score in the range of 7-15 (to minimize including subjects with knee OA so severe they may be better served by arthroplasty)
4. PHQ-9 scores 1-9, with at least one of the cardinal symptoms of depression (low mood or anhedonia) endorsed.
5. Modified Mini Mental State (3MS) Examination >/= 80.
6. Has or is willing to establish care with a personal physician prior to any experimental procedures.

Exclusion Criteria:

1. Major Depressive Episode or anxiety disorder within the past 1 year
2. Currently taking an antidepressant
3. History of bipolar or schizophrenia
4. Drug or alcohol use disorder within the past 12 months
5. Receiving knee-related workers compensation or involved in knee pain-related litigation.
6. Currently taking an anti-anxiety medicine > 4 times/week for the past 4 weeks.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change for Knee Pain | Assessed after the 8-16 week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jordan F Karp, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Late Life Depression Program, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Collins LM, Murphy SA, Strecher V. The multiphase optimization strategy (MOST) and the sequential multiple assignment randomized trial (SMART): new methods for more potent eHealth interventions. Am J Prev Med. 2007 May;32(5 Suppl):S112-8. doi: 10.1016/j.amepre.2007.01.022. PMID 17466815
- [Background] Beissner K, Henderson CR Jr, Papaleontiou M, Olkhovskaya Y, Wigglesworth J, Reid MC. Physical therapists' use of cognitive-behavioral therapy for older adults with chronic pain: a nationwide survey. Phys Ther. 2009 May;89(5):456-69. doi: 10.2522/ptj.20080163. Epub 2009 Mar 6. PMID 19270046
- [Derived] Karp JF, Zhang J, Wahed AS, Anderson S, Dew MA, Fitzgerald GK, Weiner DK, Albert S, Gildengers A, Butters M, Reynolds CF 3rd. Improving Patient Reported Outcomes and Preventing Depression and Anxiety in Older Adults With Knee Osteoarthritis: Results of a Sequenced Multiple Assignment Randomized Trial (SMART) Study. Am J Geriatr Psychiatry. 2019 Oct;27(10):1035-1045. doi: 10.1016/j.jagp.2019.03.011. Epub 2019 Mar 21. PMID 31047790
- See also: University of Pittsburgh Institute on Aging — http://www.aging.pitt.edu/
- See also: Late-Life Depression Treatment and Prevention Center at the University of Pittsburgh — http://www.wpic.pitt.edu/research/depr/
- See also: Description of clinical trial for older adults with low back pain and depression — http://www.ADAPTstudy.com